CLINICAL TRIAL: NCT03903237
Title: Herpes Zoster: Risk Factors, Complications and Special Situations- a Retrospective Analysis
Brief Title: Herpes Zoster: Risk Factors, Complications and Special Situations
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02270; sp19Mueller2
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Herpes Zoster
Keywords: post-zoster neuralgia; Herpes Zoster-related complications
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective chart review — retrospective report review of HZ patients treated between 2005 and 2018 in the Department of Dermatology at the University Hospital Basel

SUMMARY:
This retrospective analysis is to investigate patients' history and clinical presentation in Herpes Zoster (HZ), Zoster-related complications, post-Zoster neuralgia and Herpes Zoster management in order to improve the management of HZ patients, to refine HZ-vaccination strategies and elucidate cost factors of HZ in in the setting of a university hospital in Switzerland generally and in a dermatology department specifically.

ELIGIBILITY:
Inclusion Criteria:

* Reports of patients with HZ at University Hospital Basel between 2004-2018

Exclusion Criteria:

* rejection to use patient data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with HZ who were seen at University Hospital Basel between 2004-2018
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of patients' history | single time point assessment at baseline
  Free text evaluation of patients' history (age, sex, comorbidities, immunosuppression, obesity, human immune deficiency Virus (HIV), profession, current medication, vaccinations, seasonal occurence of HZ, history of Varicella Zoster virus (VZV) infection
Description of the clinical presentation of HZ | single time point assessment at baseline
  Free text description of the clinical presentation of HZ (localisation, dermatomes affected), Zoster-related acute pain
Evaluation of zoster-related complications | single time point assessment at baseline
  Free text evaluation of zoster-related complications (ophthalmic zoster, generalised HZ, Ramsay-Hunt syndrome, zoster meningoencephalitis)
Evaluation of the herpes zoster management | single time point assessment at baseline
  Free text evaluation of the herpes zoster management (local (antiviral) treatment, systemic antiviral and other treatments, number of revisits, average treatment-related costs, hospitalisations (rate, duration)
Assessment of post-zoster neuralgia | single time point assessment at baseline
  Free text assessment of post-zoster neuralgia (annual incidence, treatment options used)
Evaluation of zoster and pregnancy | single time point assessment at baseline
  Free text evaluation of zoster and pregnancy (incidence, time of pregnancy, pregnancy outcomes and complications)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Müller, Dr. med, Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland